CLINICAL TRIAL: NCT00252993
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of DDP225 in Patients With Chronic Functional Vomiting
Brief Title: 12 Weeks Treatment With DDP225 or Placebo in Patients With Chronic Functional Vomiting
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Dynogen Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DDP225-04-005
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Vomiting
Keywords: Nausea; Vomiting; Chronic Functional Vomiting; Functional Vomiting; Cyclic Vomiting
MeSH Terms: conditions — Vomiting; Nausea

INTERVENTIONS:
Drug: DDP225

SUMMARY:
This is a randomized, double blind, placebo controlled, multicenter study designed to assess the safety and efficacy of DDP225 in patients with chronic functional vomiting. Male or female patients from 18 to 65 years of age with a functional vomiting history for at least 12 weeks in the preceding 12 months or cyclic vomiting history with at least 3 episodes in the previous 12 months are eligible. A total of 30 eligible patients with chronic functional vomiting will be enrolled.

The total duration of study participation for an individual patient is approximately 15 weeks (105 days) from the initial screening visit to final study evaluations. The total duration of dosing with study medication (either DDP225 or placebo) is 12 weeks.

Patients who satisfy all of the inclusion criteria and none of the exclusion criteria are eligible to enter the Treatment Period and will be randomly assigned to one of three treatment groups.

After a patient is randomized and enters the Treatment Period, he/she will take the appropriate study medication once a day for 84 days and return to the clinic at two week intervals for a total of six visits during the Treatment Period. During the Treatment Period, patients will maintain a daily diary and complete questionnaires. One week after completing the 84-day Treatment Period, patients return to the clinic for final safety evaluations which include a physical examination, electrocardiogram, and clinical laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients from 18 to 65 years of age, inclusive.
2. History of functional vomiting for at least 12 weeks (which need not be consecutive) in the preceding 12 months, or history of cyclic vomiting with at least 3 episodes in the previous 12 months.
3. Female patients must have negative serum and urine pregnancy tests and be post-partum for at least one year or not breast feeding at the initial screening visit and throughout the study. For female patients able to bear children, an acceptable method of birth control must be used throughout the study. Patients unable to bear children must have documentation of such in the case report form (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
4. Able to provide voluntary, written informed consent with full comprehension of all aspects of the protocol.

Exclusion Criteria:

1. Serious underlying diseases (cardiovascular, genitourinary, urinary, thyroid or hematological diseases, psychiatric disorders, central nervous system disorders, or coagulation disorders).
2. Clinically significant abnormal examination findings or laboratory tests.
3. Inability to stop taking certain medications, or a planned change in medication (including herbal remedies) which would interfere with study assessments.
4. Use of drugs or ethanol which may interfere with compliance of study procedures or influence study outcome.
5. Presence of a medical condition which could interfere with the interpretation of study data.
6. Significant use of nicotine or caffeine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-11; Study Completion 2006-03

PRIMARY OUTCOMES:
Frequency and intensity of nausea and vomiting episodes

SECONDARY OUTCOMES:
Patient reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ray Clouse, MD, Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (6):
  - University of South Alabama, Mobile, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri